CLINICAL TRIAL: NCT00828386
Title: A Randomized, Multicenter, Phase III Trial Comparing Induction CT With Docetaxel, Cisplatin and 5-FU (TPF) Followed by Concurrent CT-RT to Concurrent CT Alone, in Nasopharyngeal Cancers Staged as T2b, T3, T4 and/or With Lymph Node Involvement (>N1)
Brief Title: Induction Chemotherapy and Chemoradiotherapy in Nasopharyngeal Cancers
Acronym: NPC2006
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Low accrual
Sponsor: Groupe Oncologie Radiotherapie Tete et Cou (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GORTEC NPC2006
Record Dates: First submitted 2009-01-22; First posted 2009-01-23 (Estimated); Last update posted 2019-01-18 (Actual); Status verified 2019-01

CONDITIONS: Nasopharyngeal Cancers
Keywords: Nasopharyngeal cancers; induction chemotherapy; radiochemotherapy
MeSH Terms: conditions — Nasopharyngeal Neoplasms | interventions — Induction Chemotherapy

ARMS (2):
- Induction chemotherapy + concurrent chemoradiotherapy (Experimental): Induction chemotherapy (Docetaxel + Cisplatin + 5-FU):
  * Docetaxel 75 mg/m² administered on D1 of each course, every 3 weeks, via one-hour IV infusion
  * Cisplatin 75 mg/m² administered on D1 via one-hour infusion followed by
  * 5-Fluorouracil (as a continuous infusion): 750 mg/m²/d administered as a continuous infusion from D1 to D5.
  The cycles will be repeated every 3 weeks up to a total of 3 courses. Followed by concurrent chemoradiotherapy with Cisplatin : weekly Cisplatin 40 mg/m2 starting on D1 of the radiation therapy (70 Gy/7 weeks).
  Interventions: Procedure: Induction chemotherapy + concurrent radiochemotherapy vs. concurrent radiochemotherapy
- Concurrent radiochemotherapy alone (Active Comparator): Concurrent chemoradiotherapy with Cisplatin : weekly Cisplatin 40 mg/m2 starting on D1 of the radiation therapy (70 Gy/7 weeks).
  Interventions: Procedure: Induction chemotherapy + concurrent radiochemotherapy vs. concurrent radiochemotherapy

INTERVENTIONS:
Procedure: Induction chemotherapy + concurrent radiochemotherapy vs. concurrent radiochemotherapy — Induction chemotherapy (Docetaxel, Cisplatin and 5-Fluorouracil) + concurrent radiochemotherapy

SUMMARY:
This is a randomized, multicenter, phase III trial comparing induction chemotherapy with Docetaxel, Cisplatin and 5-Fluorouracil (TPF) followed by concurrent chemoradiotherapy to concurrent chemoradiotherapy alone, in nasopharyngeal cancers staged as T2b, T3, T4 and/or with lymph node involvement (≥ N1. The main end point is the event free survival.

DETAILED DESCRIPTION:
This is a randomized, multicenter, phase III trial comparing induction chemotherapy with Docetaxel, Cisplatin and 5-Fluorouracil (TPF) followed by concurrent chemoradiotherapy (Arm A) to concurrent chemoradiotherapy alone (Arm B), in nasopharyngeal cancers staged as T2b, T3, T4 and/or with lymph node involvement (≥ N1. The main end point is the event free survival.

The treatments are :

Arm A:

induction chemotherapy: Docetaxel (75 mg/m² administered on D1 of each course, every 3 weeks via one-hour IV infusion) + Cisplatin(75 mg/m² administered on D1 via one-hour infusion )+ 5-FU (750 mg/m²/d administered as a continuous infusion from D1 to D5. The cycles will be repeated every 3 weeks up to a total of 3 courses.

followed by chemoradiotherapy with Cisplatin (40 mg/m2 starting on D1 of the radiation therapy) during 7 weeks

Arm B: Chemoradiotherapy with Cisplatin alone (40 mg/m2 starting on D1 of the radiation therapy) during 7 weeks

ELIGIBILITY:
Inclusion Criteria:

1. WHO II-III carcinoma of the nasopharynx, histologically proven by a nasal cavity biopsy, locally advanced T2b, T3, T4 and/or N1, N2 or N3 (UICC/AJCC2002).
2. Absence of distant metastases, confirmed by a chest CT scan, abdominal ultrasound (or CT scan) in case of abnormal hepatic function, and bone scintigraphy required.
3. Total absence of previous chemotherapy or radiotherapy, for whatever reason.
4. Total absence of surgical procedures for nasopharyngeal carcinoma.
5. Total absence of concurrent cancer treatment.
6. Total absence of chronic treatment (>= 3 months) with corticosteroids with a daily dosage >= 20 mg/day of methylprednisolone or equivalent.
7. Age between 18 and 70 years.
8. Performance status 0 or 1 according to the WHO criteria.
9. Hematological function parameters performed within 10 days before inclusion:

   * Neutrophils >= 1.5 * 109/l
   * Platelets: >= 100 * 109/l
   * Hemoglobin: >= 10 g/dl
10. Hepatic function parameters performed within 10 days before inclusion:

    * Total bilirubin is normal
    * AST (SGOT) and ALT (SGPT) <= 2.5 * upper limit of normal (ULN) of each center.
    * Alkaline phosphatase <= 2.5 * ULN.
11. Renal function parameters performed within 10 days before inclusion: Creatinine clearance must be <= 55 ml/min.
12. Patient who has given his/her written consent before any specific procedure of the protocol.
13. Patient having a Social Security (social policy-holders)

Exclusion Criteria:

1. WHO I carcinoma of the nasopharynx, histologically proven by a nasal cavity biopsy.
2. Other previous or concomitant cancer, except for in situ cervical cancer and cutaneous basal cell carcinoma.
3. Histological diagnosis on a lymph node biopsy.
4. Pregnant or breast-feeding females, or females and males of childbearing potential not taking adequate contraceptive measures.
5. Symptomatic peripheral neuropathy with grade >= 2 according to the NCI-CTC criteria.
6. Other serious concurrent medical disease (non-exhaustive list):

   * Unstable heart disease despite treatment.
   * Myocardial infarction within 6 months before inclusion in the trial.
   * A history of neurological or psychiatric events such as dementia, convulsions.
   * Severe uncontrolled infection.
   * Active gastroduodenal ulcer.
   * Obstructive Pulmonary Disease requiring hospitalization within the year prior to inclusion.
7. Clinical impairment of auditory function.
8. The presence, at time of screening, of psychological, familial, social or geographical factors that may have an effect on the compliance of the patient with the study protocol and monitoring comprises an exclusion criterion. These factors must be discussed with the patient before his or her inclusion in the trial.
9. Hypersensitivity to the excipients.
10. A patient already enrolled in another therapeutic trial on an investigational compound.
11. A person deprived of liberty or in the care of a guardian.

    -

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 83 (Actual)
Dates: Start 2009-01; Primary Completion 2017-04-19 (Actual); Study Completion 2017-04-19 (Actual)

PRIMARY OUTCOMES:
Event free-survival | 3 years

SECONDARY OUTCOMES:
Survival | 3 years
late and acute toxicity according to NCI-CTC and EORTC/RTOG criteria | early and late
Cumulative incidence of loco-regional progression | 3 years
Cumulative rate of metastasis | 3 years
Global response to chemo-radiotherapy | 3 years
Global response to induction chemotherapy | after the induction chemotherapy of the last patient included

CONTACTS AND LOCATIONS:
Overall Officials: Jamel Daoud, Pr, Principal Investigator — Hôpital Habib Bourguiba-3029 Sfax-Tunisie; Mounir FRIKHA, Pr, Principal Investigator — Hôpital Habib Bourguiba-3029 Sfax-Tunisie; Jean BOURHIS, Pr, Principal Investigator — Institut Gustave Roussy, 39 rue Camille Desmoulin, Villejuif, France
Locations (5):
- France (2):
  - Hôpital de la Pitié-Salpétrière, Paris
  - Institut Gustave Roussy, Villejuif
- University of Casablanca, Casablanca, Morocco
- University of Cluj, Cluj-Napoca, Romania
- Hôpital Habib Bourguiba, Sfax, Tunisia

REFERENCES:
- [Derived] Tao Y, Auperin A, Graff P, Lapeyre M, Gregoire V, Maingon P, Geoffrois L, Verrelle P, Calais G, Gery B, Martin L, Alfonsi M, Deprez P, Bardet E, Pignon T, Rives M, Sire C, Bourhis J. Very accelerated radiotherapy or concurrent chemoradiotherapy for N3 head and neck squamous cell carcinoma: Pooled analysis of two GORTEC randomized trials. Oral Oncol. 2017 Aug;71:61-66. doi: 10.1016/j.oraloncology.2017.06.002. Epub 2017 Jun 9. PMID 28688693
- [Derived] Bourhis J, Sire C, Graff P, Gregoire V, Maingon P, Calais G, Gery B, Martin L, Alfonsi M, Desprez P, Pignon T, Bardet E, Rives M, Geoffrois L, Daly-Schveitzer N, Sen S, Tuchais C, Dupuis O, Guerif S, Lapeyre M, Favrel V, Hamoir M, Lusinchi A, Temam S, Pinna A, Tao YG, Blanchard P, Auperin A. Concomitant chemoradiotherapy versus acceleration of radiotherapy with or without concomitant chemotherapy in locally advanced head and neck carcinoma (GORTEC 99-02): an open-label phase 3 randomised trial. Lancet Oncol. 2012 Feb;13(2):145-53. doi: 10.1016/S1470-2045(11)70346-1. Epub 2012 Jan 18. PMID 22261362